CLINICAL TRIAL: NCT02363478
Title: Long Term Effect of Buspirone on Esophageal Function and Esophageal Symptoms in Patients With Systematic Sclerosis (SSc)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Laikο General Hospital, Athens (Other)
Responsible Party: Principal Investigator, Assist. Profesor George Karamanolis, Assistant Professor in Gastroenterology, Laikο General Hospital, Athens
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Laikon 181/21-02-2014
Record Dates: First submitted 2015-01-29; First posted 2015-02-16 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-08

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Buspirone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- buspirone (Experimental): 4-weeks buspirone administration (20mg) in patients with SSc and esophageal involvement
  Interventions: Drug: buspirone

INTERVENTIONS:
Drug: buspirone — buspirone 10 mg X2 for 4 weeks
  Other Names: bespar

SUMMARY:
Esophagus is commonly affected in Systemic Sclerosis (SSc) and esophageal function is compromised in about 75% of patients. Previous studies have shown that buspirone, an orally available 5-HT1A (serotonin 1a receptor agonist), enhances esophageal motility in healthy volunteers. Recently, the investigators observed that a single dose of buspirone (10mg) improves lower esophageal sphincter (LES) function in patients with SSc and esophageal involvement .

Objectives: To evaluate the effect of continuous administration of buspirone on esophageal dysfunction and related symptoms in SSc using high resolution manometry (HRM).

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a chronic autoimmune disease affecting the skin and other organs especially the gastrointestinal tract. Esophageal involvement occurs in up to 90% of SSc patients. Symptoms of esophageal disease are due to gastroesophageal reflux disease (GERD) and esophageal motor dysfunction. Thus, heartburn, regurgitation and dysphagia have been reported by 80% of SSc patients.

The gold standard method for the assessment and detection of esophageal dysmotility in SSc patients is manometry. High-resolution manometry (HRM) is the most accurate tool to assess esophageal motility using multiple closely spaced (<2cm) pressure sensors, assessment of esophageal motility is more sensitive ,and allows a better assessment of LES and of the whole esophagus.

Buspirone, an orally available 5-HT1A receptor agonist, exerts a beneficial acute effect on esophageal motor dysfunction and LES pressure and may enhances an important role in improvement of esophageal symptoms in SSc patients. Thus, the investigators will conduct a study to evaluate the putative beneficial long-term effect of buspirone i) on esophageal motor dysfunction and ii) on esophageal symptoms in symptomatic SSc patients.

ELIGIBILITY:
Inclusion Criteria:

* SSc patients with esophageal symptoms

Exclusion Criteria:

* none

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Karamanolis, Principal Investigator — Academic Department of Gastroenterology, Laikon GH
Locations (1):
- Academic Department of Gastroenterology, Laikon GH, Athens, Greece

REFERENCES:
- [Derived] Karamanolis GP, Panopoulos S, Denaxas K, Karlaftis A, Zorbala A, Kamberoglou D, Ladas SD, Sfikakis PP. The 5-HT1A receptor agonist buspirone improves esophageal motor function and symptoms in systemic sclerosis: a 4-week, open-label trial. Arthritis Res Ther. 2016 Sep 1;18(1):195. doi: 10.1186/s13075-016-1094-y. PMID 27586891

RESULTS

PARTICIPANT FLOW:
Groups:
- Buspirone: Participants received buspirone 20 mg/day for 4 weeks
Period: Overall Study
Arm/Group | Buspirone
Started | 30
Completed | 22
Not Completed | 8
Not completed — Lost to Follow-up | 4
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Groups:
- Buspirone: 22 out of 30 participants (19 female) completed the study.
Arm/Group | Buspirone
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 3
Region of Enrollment [Number; unit: participants]
  Greece | 22

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline in Manometric Parameters: i) Amplitude of Contractions at the Distal Part of the Esophagus and ii) Resting and Residual (Lower Esophageal Pressure) LES Pressure and IRP (Integrated Relaxation Pressure) at Week 4
Time Frame: before and after 4 weeks buspirone administration
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Buspirone
Number analyzed (Participants) | 22
mmHg
  amplitude | 0.9 (0.2)
  LES resting pressure | 4.5 (0.7)
  LES residual pressure | 0.3 (0.2)
  IRP | 0.4 (0.2)
Statistical Analysis 1: Comparison: Buspirone; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; This statistical analysis applies to changes of amplitude of contractions, resting LES pressure and IRP between baseline and week 4

2. Primary Outcome: Changes From Baseline in Manometric Parameters: Duration of Contractions at the Distal Part of the Esophagus at Week 4
Time Frame: before and after 4 weeks buspirone administration
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Buspirone
Number analyzed (Participants) | 22
sec | 0.5 (0.4)

3. Primary Outcome: Changes From Baseline in Manometric Parameters: Velocity of Contractions at the Distal Part of the Esophagus at Week 4
Time Frame: before and after 4 weeks buspirone administration
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Buspirone
Number analyzed (Participants) | 22
cm/sec | 0.3 (0.5)

4. Secondary Outcome: Changes in the Severity of Esophageal Symptoms at Week 4
Description: Severity of esophageal symptoms (dysphagia, heartburn, regurgitation and chest pain) was measured on a 100-point visual analogue scale (VAS) ranging from 0 (absent) to 100 (very severe). Even minor decrease in the VAS score for each symptom at week 4 considered as improvement.
Time Frame: before and after 4 weeks buspirone administration
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buspirone
Number analyzed (Participants) | 22
units on a scale
  heartburn | 14.9 (7.8)
  regurgitation | 13.2 (2.7)
  dysphagia | 6.9 (8.8)
  chest pain | 1.9 (3.1)
Statistical Analysis 1: Comparison: Buspirone; Test type: Superiority or Other; p = 0.05, t-test, 2 sided; This statistical analysis applies to changes of amplitude of heartburn, regurgitation, chest pain and dysphagia between baseline and week 4

ADVERSE EVENTS:
Groups:
- Buspirone: Participants received bouspirone 20 mg/day for 4 weeks
Arm/Group | Buspirone
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 4/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Buspirone (N=30)
dizziness (Ear and labyrinth disorders) | 2
nausea (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes